CLINICAL TRIAL: NCT04796129
Title: Evaluation of the Correlation of the Inflammatory Parameters With Pain and Radiological Findings in Patients With Coxarthrosis
Brief Title: Correlation of the Inflammatory Parameters With Pain and Radiological Findings in Coxarthrosis
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: Kanuni Sultan Suleyman Training and Research Hospital (Other); Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Merve Damla Korkmaz, Principle investigator, Istanbul University
Other Study IDs: 2020/329
Record Dates: First submitted 2021-02-10; First posted 2021-03-12 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis, Hip; Inflammation; Pain
Keywords: hip osteoarthritis; inflammation; pain severity; pain level
MeSH Terms: conditions — Osteoarthritis, Hip; Inflammation; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with hip osteoarthritis: the patients who aged 45 and older and have paint in the hips. and also without having any other comorbidities about inflammatory status.
  Interventions: Other: the patients with hip osteoarthritis and their inflammatory status
- control: the participants who have any other comorbidities for impact on the inflammatory status and also no hip pain.
  Interventions: Other: the patients with hip osteoarthritis and their inflammatory status

INTERVENTIONS:
Other: the patients with hip osteoarthritis and their inflammatory status — The participants in the experimental group will be evaluated for the hip osteoarthritis. They will take and X-ray for hip joints and also hemogram for the excluding the inflammatory diseases.

SUMMARY:
Osteoarthritis (OA) is a functional disease with joint degeneration with subchondral and periosteal lesions. Coxarthrosis (or hip osteoarthritis) is an important cause of disability, especially in the advanced age group.Although hip osteoarthritis is often thought to be a non-inflammatory pathology, recent studies have shown that joint degeneration is correlated with the production of inflammatory factors and cartilage destroying enzymes.

There are very few studies evaluating the correlation of Neutrophil lymphocyte ratio, monocyte lymphocyte ratio and Platelet lymphocyte ratio with inflammatory parameters CRP and ESR levels in hip osteoarthritis and its relation with the staging of hip osteoatritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a disease characterized by joint degeneration with subchondral and periosteal lesions . Coxarthrosis (hip osteoarthritis) is an important cause of disability, especially in the advanced age group. The risk of symptomatic coxarthrosis in persons up to the age of 85 is approximately 25%. There is a possibility of total hip replacement at a rate of approximately 10% due to advanced stage coxarthrosis. Kellgren-Lawrence staging system is used to show disease severity in osteoarthritis staging. According to this, Stage 0: there is no radiological change, Stage 1: there is a slight narrowing in the joint space, Stage 2: osteophytes are formed in the joint space with stenosis in the anteroposterior radiography, Stage 3: multiple osteophytes, significant narrowing of the joint space, sclerosis and Stage 4 It describes a situation accompanied by large osteophytes, severe stenosis in the joint space, prominent sclerosis, and bone deformities.

Although coxarthrosis is often thought to be a non-inflammatory pathology, recent studies have shown that joint degeneration correlates with the production of inflammatory factors and cartilage destroying enzymes. At the cellular level, it has been found that macrophage and perivascular T and B lymphocyte infiltration play a role in early and advanced stage OA.

Neutrophils and lymphocytes are the main determinants of the inflammatory process. The neutrophil to lymphocyte ratio (NLR) is obtained by dividing the absolute neutrophil count by the number of lymphocytes obtained from the peripheral blood count. They are used as an indicator of the inflammatory process in inflammatory conditions such as ankylosing spondylitis, sarcoidosis, and cancers. In addition, platelet lymphocyte ratio (PLR) has also been found to be associated with disease activity and severity in diseases such as rheumatoid arthritis and psoriatic arthritis. Its use in the diagnosis and follow-up of OA has not yet been clearly demonstrated. However, changes in mean platelet volume are also used as an indicator of disease severity in systemic inflammatory diseases.

There are very few studies evaluating the correlation of Neutrophil lymphocyte ratio, monocyte lymphocyte ratio and Platelet lymphocyte ratio with inflammatory parameters CRP and ESR levels in hip osteoarthritis and its relation with the staging of hip osteoatritis. The aim of this study to evaluate of the correlation of the inflammatory parameters with pain and radiological findings in the patients with coxarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with hip osteoarthritis
* Being aged at 45 years or older

Exclusion Criteria:

* Not accept being participation in the study.
* Having any systemic disease like the diabetes mellitus, hypertension, coronary after disease
* Having any inflammatory rheumatologic disease
* Having any disease that prevent to participate the study like mental retardation, dementia and psychotic disorders.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the participants in the experimental group are at aged 45 years or older and have hip osteoarthritis the participants in the control group are at aged 45 years or older and have no any other diseases that effect the inflammatory status
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 day
  pain of the hip joints of the participants. It will be evaluated by using Visual Analog Scale(VAS). The scale is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations. The pain range is from 1 to 10. The minimum value is 1 and it means the pain is so mild. The maximum value is 10, it means the pain is so much, like a knife stabs.
NLR | 1day
  neutrophil lymphocyte ratio
PLR | 1 day
  platelet lymphocyte ratio
MLR | 1 day
  monocyte lymphocyte ratio
ESR | 1 day
  Erythrocyte Sedimentation Ratio
CRP | 1 day
  C-reactive protein
X-ray of hip joints | 1 day
  an AP X-ray for the painful hip joints
Lequesne Index | 1 day
  pain severity

CONTACTS AND LOCATIONS:
Overall Officials: Merve Damla Korkmaz, 1, Principal Investigator — Istanbul University
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication)
Supporting Information: Study Protocol
Time Frame: The data will be available after publication
Access Criteria: The data will share with permission and request.